CLINICAL TRIAL: NCT02014948
Title: Implementation of a Physiotherapy Intervention for Patients With Chronic Low Back Pain
Brief Title: Vibratory Therapy for Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratório de Engenharia de Reabilitação Sensorio Motora (Other)
Responsible Party: Principal Investigator, Djenifer Queiroz de Souza, Djenifer Queiroz de Souza, Laboratório de Engenharia de Reabilitação Sensorio Motora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 13527313.3.0000.5503
Record Dates: First submitted 2013-11-07; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Physiotherapy
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercises (Experimental): This group will consist of 20 individuals, 10 with lumbar disc herniation and 10 with chronic low back pain who underwent treatment with exerxises.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — The individuals who make up this group performed exercises for 10 consecutive sessions.

SUMMARY:
The lumbar spine is currently one of the most affected areas by nociceptive processes , referred back pain, which can be provided from a herniated intervertebral disc . Such conditions are considered a public health problem , since considerably affect the population , mainly young adults , which may lead to functional disability and absenteeism . Soon , his treatment involves high costs and rehabilitation time indefinite , generating great scientific interest focused on the search for new techniques that can provide an acceleration of functional recovery of these individuals .

Thus , the establishment of evaluation protocols that provide quantitative data concerning the functional capacity is of utmost importance . From the electromyographic analysis , one can measure the electrical activity of muscle and identify abnormal patterns of response. For the identification of kinematic changes becomes useful equipment capable of recording the speed and angle of movement, as the accelerometer . Another evaluation method applicable to cases of herniated disc and back pain is the force platform to quantify the ground reaction force during the stance phase of the movement . Also , the quality of life should be taken into account as routinely observed psychological impairment involving issues related to vitality, emotional and social aspects , which can be identified through the questionnaire of quality of life ( SF -36 ) .

With regard to physical therapy intervention , we seek to use resources to compose promising treatment program along with conventionalexercises. A novel therapy in the treatment of back pain is the whole body vibration , as it promotes increased range of muscle spindles via increasing the tonic vibration reflex and consequently improving the mechanism of involuntary muscle control . Thus , the association between an accurate assessment , exercises and therapy vibratory seeks early rehabilitate individuals affected by back pain or herniated disc , delaying or even avoiding surgery .

DETAILED DESCRIPTION:
There are currently various treatment techniques have been employed for the rehabilitation of patients with functional back pain in general. However , it is essential to search for resources to compose the therapeutic treatment program along with conventional exercises.

With regard to the functional rehabilitation , physical therapy , has emphasized the muscles directly involved in the painful process (Richardson et al . , 1999) . Through exercises primarily used in functional rehabilitation , it is possible to treat and prevent impairments , restore function , promote physical and social well being . The therapeutic approach of the column follows the same principles as other structures , keeping up the proper precautions concerning the region's proximity to the spinal cord and nerve roots ( Kisner , Colby , 2005) . On this basis several treatments have been proposed , however , the most effective therapy is still a matter of controversy .

It is known that back pain can result in neurological imbalances , mainly affecting the deep muscles of the trunk and paraspinal , multifidus and transversus abdominis ( LINDGREN et al . , 1993; HIDES ; Richardson , Jull , 1996; HODGES ; Richardson , Jull , 1996). We observe a reduction in these shooting action potential and changes in motor control , represented by weakness, atrophy and reduced functional capacity ( HODGES ; MOSELEY , 2003; MACDONALD ; MOSELEY ; HODGES , 2006; RENKAWITZ ; BOLUKI ; Grifka , 2006 , RICHARDSON ; HODGES ; HIDES , 2004; BARR ; GRIGGS ; Cadby , 2007) .

Therefore, an appropriate exercise program should be able to provide muscular support , minimizing the risk of disability by recovering the functionality of the spine ( McFeely ; GRACEY , 2006). For this purpose it is recommended to strengthen the abdominal muscles , lower back and lower limbs ( HANDA et al . , 2000; CALMELS et al . , 2004; Lidder ; BAXTER ; GRACEY , 2004; HAYDEN et al . , 2005; McFeely ; GRACEY , 2006; RODACKI et al . , 2008) .

Currently the lumbar stabilization is considered a beneficial technique in the treatment of patients with low back pain , because in addition to reduce painful symptoms , promotes strengthening the stabilizing muscles such as multifidus and transversus abdominis . ( O'Sullivan , TWOMEY ; Allison 1997, Richardson et al. 1999; HIDES ; jull ; Richardson , 2001; YILMAZ et al. 2,003 ; Choi et al. 2005).

In studies carried out by Kjellby - Wendt et al. (2001) , Mannion et al. (2007) Johansson et al. (2009 ) it was possible to prove that the lumbar stabilization associated with stretching and strengthening exercises for the lower back , abdominal and lower limbs was effective in reduction of pain of the patients concerned .

Furthermore, there was a close relationship of low back pain with decreased range of motion and flexibility ( Takala , 2000) . Thus , another approach indispensable and complementary treatment for herniated disc is muscle stretching , it is able to provide a reduction in pain and decreased pressure within the core ( KUUKKANEN ; Malkia , 2000; HAKKINEN et al. 2,005 ; Kisner , Colby , 2005) .

The vibration is considered an innovative feature in the treatment of chronic low back pain and herniated disc as many musculoskeletal effects are noticed from this . According to Silva (2011) for exposure to vibration, it is possible that the muscles produce a force about 15 times higher than that produced in normal conditions, in order to oppose the action of gravitational force . Cardinale and Bosco (2003 ) stated that the vibration causes changes in muscle length , so in an attempt to mitigate this effect , the afferent influence the motor response , causing modulation of muscle stiffness . According to Bishop cited Barbosa (2009 ) in response to stimulation of the muscle spindle is an isometric contraction known as the tonic vibration reflex ( RTV ) , which is accompanied by a reciprocal inhibition of the antagonist and blocking myotatic reflex .

Thus , along with the voluntary contraction , this therapy provides improved motor control and strengthening exercises , to increase the range of activation of muscle spindles triggering the tonic vibration reflex ( BOSCO ; CARDINALE ; TSARPELA , 1999; Rittweger ; BELLER ; Felsenberg , 2003; Curry ; Clelland cited DIEEN ; SELEN ; CHOLEWICHI , 2003; SILVA ; Couto ; SZMUCHROWSKI , 2008) . For present inability to generate muscle strength needed to avoid instabilities in the affected segments , the vibration becomes a relevant resource in the treatment for chronic low back pain and disc herniation ( YILMAZ et al . , 2003) .

Although they represent a major cause of pain and functional disability , does not observe the use of biomedical instrumentation for quantitative analysis in clinical practice , such as guiding therapeutic management.

For the establishment of an appropriate physical therapy intervention becomes necessary to use equipment to assess that provide quantitative data regarding the patient's functional capacity , since the current legislation does not allow the physiotherapist to request tests such as MRI , CT and rays -X. It is believed that the association between an accurate assessment and appropriate treatment can guide the therapeutic making it more effective in attenuation of pain , allowing functional improvement of patients with disc herniation and low back pain in general.

- Surface Electromyography

As a result of the pain , it triggered a defense mechanism that results in a change in motor recruitment deficit represented by the generation of muscle strength and increased agonist antagonist activation ( DIEEN ; SELEN ; CHOLEWICHI , 2003; Larivière et al . , 2003; BASSANI et al . , 2008) . Aimed at quantifying motor function becomes useful a resource as surface electromyography , which enables the recording of muscle electrical activity in real time , allowing the identification of abnormal patterns of response ( Portney , 2004) . The device comprises electrodes reference surface and connected to the unit via cables sealed , and sensor preamplifiers information leading to electrical activity , and also biofeedback unit . The collected data are stored in the computer for further analysis , normally made by means of the square root of the mean square value (RMS ) comprising the result of the signal amplitude by means of the average power in the time interval considered , containing information about the number of motor units fired at a given motion ( Hamill , Knutzen , 1999; DE LUCA , 2002; MACHADO , 2008; O ' SULLIVAN , SCHMITZ , 2010) .

- Platform Power

Another evaluation method applicable to cases of herniated disc is the force platform that consists of two rigid surfaces interconnected by means of sensors , allowing to quantify the ground reaction force during the stance phase of the movement ( BARELA ; DUARTE , 2011) . Thus , it is of great interest because patients tend to adopt an antalgic posture , reducing the weight bearing on the limb ipsilateral to the disc herniation .

- Accelerometer

It is known that patients with low back pain may suffer biomechanical changes that directly influence kinematic and kinetic parameters . Therefore , it is appropriate to examine the speed , amplitude and angle of movement . Therapists and patients can benefit from the use of a device able to provide such data in a simple and flexible , making it easy to conduct and providing greater comfort to both. Therefore , we developed a device called accelerometer , which is composed of three parts , which are : sensor , receiver and software for data conversion on the computer .

The sensor is part of the equipment positioned in the joint under consideration. Each sensor is constituted by a microcontroller, a three-axis accelerometer and a processor network . The microcontroller communicates with the accelerometer chip through a Serial Peripheral Interface ( SPI ) . When prompted , the accelerometer chip microcontroller sends the values of X , Y and Z corresponding to the force vector ( Gaino , 2010) . From these values the microcontroller assembles a data packet to be sent via wireless communication . The processor sensor network is restricted to connecting to the network , and is therefore called end device .

The function of the receiver is receiving the sensor data and send them via serial communication to the computer . Finally , a software program is responsible for converting data received from the accelerometer sensor .

To determine the angle of inclination of a certain body part, the program is designed to break the force vector of three vectors ( X , Y, Z ) , from which one can obtain the angle of each axis if the calculation the angles of the three vectors with their respective unit vectors . The system provides the angles for the three Cartesian axes every 0.5 seconds of exercise.

The software also provides the function to calibrate , allowing to adopt the pertinent angles to each patient as a starting position , keeping the slope from this position . Data is written to a text file and automatically stored in a folder on the local disk C :/ , the identification data occurs by the date and time naming each file generated .

- Questionnaire Short Form Health Survey ( SF -36 )

Commonly , patients with chronic pain face psychological problems that directly affects their self-esteem and social interaction . Thus , we have the Short Form Health Survey ( SF -36 ) widely used in assessing the quality of life of patients with low back pain ( MILANI et al . , 2009; VERESCIAGINA ; AMBROZAITIS ; AKAUSKAS , 2009; AHRENS ; SCHILTENWOLF ; WANG , 2010; Luedtke et al . , 2011; HAUGEN et al . , 2011) . It is a non-specific questionnaire consisting of 36 items divided into social function , mental health index , physical and social function , pain index , vitality , physical appearance and emotional and general health perceptions , which concludes the evaluation protocols volunteers in this study ( Rosanova et al . , 2010) .

ELIGIBILITY:
* Inclusion criteria:

  1. Lack of diseases or complaints of back pain;
  2. Medical diagnosis of lumbar disc herniation , evidenced by imaging studies;
  3. Low back pain or sciatica in the presence of antalgic postures;
  4. 80% stake in therapy sessions;
  5. Individuals who agree to participate in this study and signed an informed consent form.
* Exclusion criteria:

  1. Presence of vertebral pathologies or symptoms that involve the same;
  2. The use of anti -inflammatory steroids or nonsteroidal;
  3. Women in menstrual period;
  4. Pregnant or postpartum;
  5. Cognitive deficits;
  6. Hyperesthesia, hypoesthesia or anesthesia evaluated muscle group;
  7. Surgery in the previous column;
  8. The presence of infiltration of corticosteroids in less than six months;
  9. The use of anti -inflammatory steroids or nonsteroidal;
  10. The use of analgesics;
  11. Cognitive deficits;
  12. Collections in menstrual period;
  13. Pregnant and postpartum;
  14. Hemorrhage;
  15. Malignancy;
  16. Diabetes mellitus;
  17. Deep venous thrombosis;
  18. Regions healing;
  19. Acute inflammation;
  20. Fracture healing;
  21. Pressure ulcers.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Electromyographic analysis of the trunk erector of patients with chronic low back pain . | Thirty seconds.
  All groups performed the evaluation of muscle electrical activity , using a surface electromyography , 2 channels ( EMG System ® ) , model EMG 230C - USB , composed of an analog-digital converter 12-bit resolution and power supply to battery to avoid interference from the power grid . The parameters used were : sampling frequency of 2,000 Hz , unit uV , -2000 Xmin , Ymax 2000 Coef . The 0 and Coef . B 500.
  The electrodes were then fixed in pairs , respecting the distance of 2 cm between them ; longitudinally over the belly of the erector muscles of the trunk . Data were collected in the prone and standing for 30 seconds , during which the subject performed the isotonic contraction muscle evaluated .

SECONDARY OUTCOMES:
Analysis of pain using a visual analogue scale . | Two days.
  The subjects were instructed to respond to a visual analogue scale with the level 0 as no pain and 10 as state level of maximum pain .

OTHER OUTCOMES:
Force Platform | Thirty seconds
  The acquisition of data on the force platform lasted 30 seconds , during which patients took the standing position in the region previously marked on the equipment , so that the support base was identical for all volunteers . Also , samples were collected at rest , followed by consecutive flexion-extension of the trunk .

CONTACTS AND LOCATIONS:
Overall Officials: Djenifer Q Souza, Therapy, Principal Investigator — University of Vale of Paraiba
Locations (1):
- University of Vale of Paraiba, São José dos Campos, São Paulo, Brazil

REFERENCES:
- [Background] Basbaum AI, Bautista DM, Scherrer G, Julius D. Cellular and molecular mechanisms of pain. Cell. 2009 Oct 16;139(2):267-84. doi: 10.1016/j.cell.2009.09.028. PMID 19837031
- [Background] AHRENS, C.; SCHILTENWOLF, M.; WANG, H. Health-related quality of life (SF-36) inchronic low back pain and comorbid depression. Schmerz, v. 24, n. 3, p. 251-256, 2010. BASSANI, E. et al. Avaliação da ativação neuromuscular em indivíduos com escoliose através da eletromiografia de superfície. Rev. bras. fisioter., v. 12, n. 1, p. 13-19, 2008. BOSCO, C.; CARDINALE, M.; TSARPELA, O. Infuence of vibration on mechanical power and electromyogram activity in human arm flexor muscles. Eur. J. Appl. Physiol., v. 79, p. 306-311, 1999. BRAZIL et al. Diagnóstico e tratamento das lombalgias e lombociatalgias. Rev. Bras. Reumatol., v. 44, n. 6, p. 419-425, 2004. KISNER, C.; COLBY, L. A. Exercícios Terapêuticos: fundamentos e técnicas. 4 ed., Barueri: Manole, 2004. LIZIER, D. T. et al. Exercícios para tratamento de lombalgia inespecífica. Rev. Bras. Anestesiol., v. 62, n. 6, p. 838-846, 2012.
- See also: The nervous system detects and interprets a wide range of stimuli. When plasticity facilitates protective reflexes , can be beneficial , but when the changes persist , a condition of chronic pain can result . — http://www.ncbi.nlm.nih.gov/pubmed?term=Basbaum+AI%5Bauthor%5D+AND+Cellular+and+Molecular+Mechanisms+of+Pain&TransSchema=title&cmd=detailssearch